CLINICAL TRIAL: NCT04678102
Title: A Phase I, Open-label, Dose-finding Study to Assess the Safety, Tolerability, and Pharmacokinetics of PHI-101 in Patients With Platinum-Resistance/Refractory Ovarian Cancer
Brief Title: Chk2 Inhibitor for Recurrent EpitheliAl periToneal, fallopIan or oVarian cancEr (CREATIVE Phase IA Trial)
Acronym: CREATIVE
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Pharos iBio Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Hee Seung Kim, Associate Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PHI-101-002
Record Dates: First submitted 2020-11-29; First posted 2020-12-21 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Platinum-resistant Ovarian Cancer; Platinum-refractory Ovarian Carcinoma; Platinum-Resistant Fallopian Tube Carcinoma; Platinum-Resistant Primary Peritoneal Carcinoma
Keywords: PHI-101; Chk2 inhibitor; antineoplastic; Platinum-resistant Ovarian Cancer
MeSH Terms: interventions — PHI-101

STUDY DESIGN:
Intervention Model Description: According to the accelerated 3+3 design, the accelerated dose escalation scheme, which assesses DLT in 1 subject in each cohort, is applied until an adverse drug reaction (ADR) ≥ [CTCAE version 5.0] grade 2 occurs. If an ADR ≥ grade 2 occurs in a specific cohort, the accelerated 3+3 design will be immediately switched to the standard 3+3 scheme, and 3 to 6 subjects will be enrolled in each cohort. If a DLT is observed in > 1 out of 6 subjects in a specific cohort (χ) and a DLT is observed in ≤ 1 out of 6 subjects in the cohort (χ-1) that is one level lower than the specific cohort, the one level lower cohort (χ-1) will be considered as the MTD. The dose of PHI-101 will be escalated until an MTD is determined. If the MTD is not determined at the MPD, dose escalation will be ended at that dose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (PHI-101 40mg/day) (Experimental): In the starting dose cohort 1 subject will be administered 40mg/day PHI-101 and will be assessed for DLT ('single subject cohort'), and until an ADR ≥ [CTCAE version 5.0] grade 2 occurs, higher doses will be explored in single subject cohorts in a stepwise fashion. If an ADR ≥ [CTCAE version 5.0] grade 2 occurs, the accelerated 3+3 design will be immediately switched to the standard 3+3 scheme.
  Interventions: Drug: PHI-101 administration
- Cohort 2 (PHI-101 80mg/day) (Experimental): In cohort 2, the subject will be administered 80mg/day PHI-101.
  Interventions: Drug: PHI-101 administration
- Cohort 3 (PHI-101 120mg/day) (Experimental): In cohort 3, the subject will be administered 120mg/day PHI-101.
  Interventions: Drug: PHI-101 administration
- Cohort 4 (PHI-101 160mg/day) (Experimental): In cohort 4, the subject will be administered 160mg/day PHI-101.
  Interventions: Drug: PHI-101 administration
- Cohort 5 (PHI-101 200mg/day) (Experimental): In cohort 5, the subject will be administered 200mg/day PHI-101.
  Interventions: Drug: PHI-101 administration
- Cohort 6 (PHI-101 240mg/day) (Experimental): In cohort 6, the subject will be administered 240mg/day PHI-101.
  Interventions: Drug: PHI-101 administration

INTERVENTIONS:
Drug: PHI-101 administration — Escalated doses of PHI-101 will be administered to each cohort.
  Other Names: PHI-101

SUMMARY:
This study aims to assess the safety and tolerability of PHI-101 in patients with platinum-resistance/refractory ovarian, fallopian tubal, and primary peritoneal cancer. This study also evaluates the pharmacokinetics of PHI-101 and efficacy of PHI-101 during treating platinum-resistance/refractory ovarian, fallopian tubal, and primary peritoneal cancer.

PHI-101 is a CHK2 inhibitor that is a checkpoint kinase binding specifically to CHK2, rather than CHK1, and it inhibits the DDR system by inhibiting the ATM-CHK2 pathway, which is activated in response to DSBs. When a high-grade serous ovarian (HGSO) cancer cell line and various ovarian cancer cell lines (CAOV3, OVCAR3, SK-OV-03, and SW626) were treated with PHI-101 in a non-clinical study, the therapeutic effect of PHI-101 against ovarian cancer was demonstrated by a decrease in viability of ovarian cancer cells. In addition, a stronger growth inhibition effect was observed compared to that of treatment with olaparib or rucaparib alone, and a much stronger inhibition effect was observed when concomitantly used with paclitaxel, cisplatin, and topotecan. Based on the aforementioned results of the non-clinical studies, the potential of PHI-101 as a new treatment or concomitant cytotoxic chemotherapeutics for patients with ovarian cancer who are resistant to existing antineoplastic drugs was confirmed.

DETAILED DESCRIPTION:
In this study, a maximum of 6 dose levels (cohorts) were planned for daily oral administration of PHI-101. Subjects who meet the inclusion/exclusion criteria of this study will be enrolled in each cohort and assessed for safety and tolerability after administering PHI-101 to determine the MTD. Subjects will be enrolled sequentially starting from the low-dose cohort, and DLT will be assessed for the first 28 days (Cycle 1) after the first dose of PHI-101. Before DLT is assessed in a specific cohort, enrolling a subsequent subject in the next higher dose cohort will not be allowed.

According to the accelerated 3+3 design, the accelerated dose escalation scheme, which assesses DLT in 1 subject in each cohort ('single subject cohort'), is applied until toxicity (ADRs) related to PHI-101 ≥ [CTCAE version 5.0] grade 2 occurs. If ADRs ≥ grade 2 do not occur in 1 subject, DLT can be assessed in one level higher cohort according to the SRC's recommendation. If an ADR ≥ grade 2 occurs in a specific cohort, the accelerated 3+3 design will be immediately switched to the standard 3+3 scheme, and 2 additional subjects will be enrolled in that cohort (1 subject + 2 additional subjects) to assess DLT during 1 cycle.

After switching to the standard 3+3 scheme, 3 to 6 subjects will be enrolled in each cohort. If no DLT is observed in the first 3 subjects, DLT can be assessed in one level higher cohort according to the SRC's recommendation. If DLT is observed in 1 out of 3 subjects (DLT: 1/3 subject), that cohort will be expanded to 6 subjects by enrolling 3 additional subjects. If 2 out of 3 to 6 subjects experience DLT (DLT: 2/3 to 6 subjects), this means that the MTD is exceeded. Thus, additional enrollment will be ended for that cohort. The one level lower cohort will expand to 6 subjects (If 6 subjects were already enrolled in that cohort, additional enrollment is unnecessary).

A subject not evaluable for DLT (withdrawal for reasons other than AEs or ADRs, or less than 20 out of 28 doses of PHI-101 were administered during Cycle 1) may be replaced by another subject according to the judgment of the investigator (decision/recommendation of the SRC, if necessary). If a subject in the single subject cohort is not evaluable for DLT, a substitute will be enrolled in the same cohort (1 subject + 1 additional subject) to assess DLT. If it is determined not to replace the subject not evaluable for DLT, the subject will be considered to have experienced DLT when the dose escalation is decided.

If DLT is observed in > 1 out of 6 subjects in a specific cohort (χ) and DLT is observed in ≤ 1 out of 6 subjects in the cohort (χ-1) that is one level lower than the specific cohort, the one level lower cohort (χ-1) will be considered as the MTD. The dose of PHI-101 will be escalated until an MTD is determined. If the MTD is not determined at the MPD, dose escalation will be ended at that dose (Addition of cohorts may be reviewed by and discussed with the SRC, if necessary, but reporting to the MFDS and the IRB and protocol amendment should occur first.) According to the schedule of activities (SOA), observation, questioning, examination, and tests to assess the safety and tolerability of PHI-101, PK sampling to assess PK, and tumor response assessment to explore efficacy will be performed.

After the EOT of PHI-101, the EOT visit will take place. Survival of subjects and initiation of new antineoplastic therapy will be periodically checked until the EOS. The follow-up will be performed for 1 year after the EOS to obtain such information.

ELIGIBILITY:
Inclusion Criteria:

1. Females aged ≥ 19 years at the time of informed consent
2. Pregnancy (childbearing potential and planning a pregnancy) and breast-feeding status ① Women of non-childbearing potential, women who are not pregnant or breast-feeding, or women who are not planning a pregnancy during the study

   ② Women of childbearing potential (Section 10.3.2.7.1) who have a confirmed negative pregnancy test at screening and immediately before administration of PHI-101 and agree to use an effective contraceptive method(s) (Section 10.3.2.7.2) required in this protocol for 6 months (24 weeks) from the last dose of PHI-101
3. Indication

   ① Histologically or cytologically confirmed ovarian cancer, fallopian tube carcinoma, or primary peritoneal cancer

   ② Epithelial malignant tumors diagnosed through local histopathological findings [WHO Histological Classification, 2014]

   : except LGSC, mucinous carcinoma of the ovary, MMMT, and LAP, which are classified as LCOH, [NCCN Guideline version 2.2019].

   LAP = low malignant potential (ovarian borderline epithelial tumor); LCOH = less common ovarian histopathology; LGSC = low-grade serous carcinoma; MMMT = malignant mixed Mullerian tumor (carcinosarcoma); NCCN Guideline = National Comprehensive Cancer Network Guideline; WHO Histological Classification = World Health Organization Histological Classification ③ Platinum-refractory cancer* or platinum-resistance cancer†
   * Disease progression during platinum-based antineoplastic therapy, † Disease progression within 6 months (24 weeks) from completion of platinum-based antineoplastic therapy ④ Inoperable subjects who are refractory to, cannot receive, or refuse standard of care, which is currently known to be clinically beneficial ⑤ Subjects with ≥ 1 measurable lesion or nonmeasurable, but evaluable lesion that meets [RECIST version 1.1] RECIST = Response Evaluation Criteria in Solid Tumors
4. Expected life expectancy ≥ 12 weeks
5. [ECOG PS] ≤ 1 ECOG PS = Eastern Cooperative Oncology Group Performance Status
6. Subjects who have adequate hepatic, renal, and hematological function confirmed by the following laboratory tests (a re-test will be allowed during the screening period) ANC ≥ 1,500/mm3 (without administration of G-CSF within 2 weeks prior to baseline) Hb ≥ 10.0 g/dL (without transfusion within 2 weeks prior to baseline) Platelet count ≥ 75,000/mm3 (without transfusion within 2 weeks prior to baseline) Total bilirubin ≤ 1.5 x ULN AST and ALT ≤ 3.0 x ULN* (≤ 5 x ULN for patients with liver metastases or hepatocellular carcinoma) Serum creatinine (or CrCl) Serum creatinine ≤ 1.5 x ULN CrCl ≥ 60 mL/min (by Cockcroft-Gault equation)
7. Prior antineoplastic therapy and treatment ① Prior cytotoxic chemotherapy ≤ 5 times

   ② Reversible side effects from prior antineoplastic therapy (operation, drug, radiation therapy, etc.)* resolved to [CTCAE version 5.0] grade 1 or better

   * Subjects should not have had major surgery, antineoplastic therapy or experimental therapy, or direct radiation therapy on hematopoietic site within 4 weeks prior to baseline and should not be administered nitrosoureas or mitomycin-C within 6 weeks prior to baseline.

   CTCAE = Common Terminology Criteria for Adverse Events
8. Subjects who voluntarily decided to participate and provided written consent after they were given sufficient explanation of this study
9. Subjects who are able to understand the study procedures and restrictions and willing to comply with them during the study

Exclusion Criteria:

* 1) Subjects with known or suspected hypersensitivity or intolerance to the active ingredient or excipients of PHI-101 2) Subjects considered ineligible or unable to participate in this study according to the investigator's judgement for other reasons

Medical history or current medical condition and disease 3) Subjects with the following cardiac insufficiency or cardiovascular disease (but not limited to):

* Evidence of myocardial ischemia or myocardial infarction within 12 weeks prior to baseline

  * [NYHA Functional Classification] ≥ II NYHA = New York Heart Association ③ LVEF < 50% confirmed by ECHO or MUGA scan LVEF = left ventricular ejection fraction; ECHO = echocardiography; MUGA = Multi-gated acquisition blood pool scintigraphy

    * Clinically significant cardiac arrhythmia that is uncontrolled by the adequate and optimal treatments

      ⑤ Corrected QT (QTc)* interval > 450 msec (for both men and women) or long QT syndrome (or family history)

      * QT interval (QTcF) corrected using Fridericia's formula will be used. In case of bundle branch block, the Bazett's formula will be used (QTcB).

      4) Subjects with the following gastrointestinal diseases that affect intake or absorption of the drug (but not limited to):
* Dysphagia

  * Paralysis of intestine and intestinal obstruction

    ③ Gastrointestinal surgery that has a clinically significant effect on absorption of the drug: gastrotomy, small intestinal fistula, extensive small bowel resection, etc. (except for simple anastomosis)

    ④ Autoimmune or inflammatory disease that involves the entire gastrointestinal system or small intestines: coeliac disease, intestinal graft versus host disease, Behcet's syndrome, scleroderma involving the gastrointestinal tract, Crohn's disease, ulcerative colitis, etc.

    5) Lung diseases (but not limited to):
* New or progressive dyspnea, cough, and fever

  ② Planned diagnosis of interstitial lung disease, or interstitial pneumonia

  ③ Pulmonary fibrosis 6) Hematologic malignancy including lymphoma 7) Metastasis:
* Central nervous system metastasis or brain metastasis ② Bone metastasis 8) Infectious disease (but not limited to):
* Severe infectious disease requiring administration of antibiotics, antivirals, etc. that may affect the safety and efficacy assessments during the study

  * Active (overt) infectious disease that is uncontrolled by the adequate and optimal treatments as determined by the investigator 9) Known positive human immunodeficiency virus (HIV) 10) Active hepatitis B* or active hepatitis C†

    * HBsAg positive with HBV DNA detected † Anti-HCV positive with HCV RNA detected (qualitatively) 11) Unintentional weight loss > 10% within 12 weeks prior to informed consent 12) History of alcohol or other drug abuse within 1 year (52 weeks) prior to informed consent

Subjects who received, are receiving, or cannot stop the following therapy (medication/non-medication) 13) Subjects who need antineoplastic therapy* other than the IP during the study participation (Point radiation to alleviate bronchial obstruction, skin lesion, etc. is allowed).

* Surgery, radio(chemo)therapy, cytotoxic chemotherapy, targeted therapy (small molecule drug, monoclonal antibody), immuno-oncology drug (biological drug), hormone therapy, etc.

14) Subjects who received (used) other investigational study product or device within 2 weeks or 5 half-lives prior to informed consent (whichever is shorter) 15) Subjects on drugs (nonprescription drug, herb, homeopathy, etc.) that have a significant effect on the assessment of kinetics (metabolism, excretion, etc. in the body) or efficacy and safety of the IP within 2 weeks prior to informed consent as determined by the investigator

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-12-17 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with dose-limiting toxicity (DLT) | Subjects will be treated and observed for DLT through the end of the first cycle (Days 1-28)
  The frequency and percentage of DLT that occurs during 1 cycle (28 days) after administration of the IP will be presented by the cohort.
Maximum tolerated dose | Through the first cycle (Day1-28)
  The dose of PHI-101 will be escalated until an MTD is determined, and if the MTD is not determined at the MPD, dose escalation will be ended at that dose

SECONDARY OUTCOMES:
Dose interruption (temporary discontinuation) percent (%) | Through the first cycle (Day1-28)
  Dose interruption percent (temporary discontinuation) of the IP due to adverse events (AEs) in each cohort will be presented using frequency and percentage, and 95% exact confidence intervals (CIs).
Dose reduction percent (%) | Through the first cycle (Day1-28)
  Dose reduction percent (%) of the IP due to adverse events (AEs) in each cohort will be presented using frequency and percentage, and 95% exact confidence intervals (CIs).
Dose termination (permanent discontinuation) percent (%) | Through the first cycle (Day1-28)
  Dose termination percent (%) of the IP due to adverse events (AEs) in each cohort will be presented using frequency and percentage, and 95% exact confidence intervals (CIs).
Cmax | Cycle1Day1, Cycle1Day8, Cycle1Day15, Cycle2Day1, Cycle3Day1, Cycle6day1, and then, every 12 weeks until end of the study, up until 24 months (each cycle is 28 days)
  Maximum plasma concentration after administration
AUCt | Cycle1Day1, Cycle1Day8, Cycle1Day15, Cycle2Day1, Cycle3Day1, Cycle6day1, and then, every 12 weeks until end of the study, up until 24 months (each cycle is 28 days)
  Area under the plasma concentration-time curve to the last measurable blood sampling time point, calculated by the trapezoidal method. AUC of the interval with increasing plasma concentration is calculated by a linear trapezoidal method, and AUC of the interval with decreasing plasma concentration is calculated by the log-linear trapezoidal summation. Concentrations below lower limit of quantification (LLOQ) will be excluded from calculation.
AUCτ | Cycle1Day1, Cycle1Day8, Cycle1Day15, Cycle2Day1, Cycle3Day1, Cycle6day1, and then, every 12 weeks until end of the study, up until 24 months (each cycle is 28 days)
  Area under the plasma concentration-time curve from time of administration to τ (AUCτ) (τ: dosing interval)
AUCinf | Cycle1Day1, Cycle1Day8, Cycle1Day15, Cycle2Day1, Cycle3Day1, Cycle6day1, and then, every 12 weeks until end of the study, up until 24 months (each cycle is 28 days)
  Area under the plasma concentration-time curve extrapolated from the time of a single dose to infinity. AUCinf = AUClast + Clast /λz
Tmax | Cycle1Day1, Cycle1Day8, Cycle1Day15, Cycle2Day1, Cycle3Day1, Cycle6day1, and then, every 12 weeks until end of the study, up until 24 months (each cycle is 28 days)
  Time to maximum plasma concentration after administration
Tmax,ss | Cycle1Day1, Cycle1Day8, Cycle1Day15, Cycle2Day1, Cycle3Day1, Cycle6day1, and then, every 12 weeks until end of the study, up until 24 months (each cycle is 28 days)
  Time to maximum plasma concentration at steady state
t1/2 | Cycle1Day1, Cycle1Day8, Cycle1Day15, Cycle2Day1, Cycle3Day1, Cycle6day1, and then, every 12 weeks until end of the study, up until 24 months (each cycle is 28 days)
  Half-life obtained by calculating ln(2)/λz, where λz is the elimination rate constant obtained from the linear regression analysis of log-linear plot at the terminal phase of the plasma concentration-time curve
PTF | Cycle1Day1, Cycle1Day8, Cycle1Day15, Cycle2Day1, Cycle3Day1, Cycle6day1, and then, every 12 weeks until end of the study, up until 24 months (each cycle is 28 days)
  Fluctuation (%) between the maximum and minimum plasma concentrations at steady state
AR | Cycle1Day1, Cycle1Day8, Cycle1Day15, Cycle2Day1, Cycle3Day1, Cycle6day1, and then, every 12 weeks until end of the study, up until 24 months (each cycle is 28 days)
  Ratio of systemic exposure of the drug at steady state to systemic exposure of the drug after a single dose
CL/F | Cycle1Day1, Cycle1Day8, Cycle1Day15, Cycle2Day1, Cycle3Day1, Cycle6day1, and then, every 12 weeks until end of the study, up until 24 months (each cycle is 28 days)
  Apparent clearance CL/F = Dose/AUCinf
CLss/F | Cycle1Day1, Cycle1Day8, Cycle1Day15, Cycle2Day1, Cycle3Day1, Cycle6day1, and then, every 12 weeks until end of the study, up until 24 months (each cycle is 28 days)
  Apparent clearance at steady state
Vdz/F | Cycle1Day1, Cycle1Day8, Cycle1Day15, Cycle2Day1, Cycle3Day1, Cycle6day1, and then, every 12 weeks until end of the study, up until 24 months (each cycle is 28 days)
  Volume of distribution in the terminal phase
Objective response rate (ORR) | Until the end of the study or death, which may be up to 24 months
  ORR = complete response (CR) + partial response (PR)
  : For subjects who have best overall response (BOR) of complete response (CR) or partial response (PR), frequency and percentage, and 95% exact CIs will be presented by cohort evaluated according to the RECIST criteria by CT imaging.
Disease control rate (DCR) | Until the end of the study or death, which may be up to 24 months
  DCR=CR+PR+SD For subjects with BOR of CR, PR, or stable disease (SD), frequency and percentage, and 95% exact CIs will be presented by cohort and evaluated according to the RECIST criteria by CT imaging.
Duration of response (DOR) | Until the end of the study or death, which may be up to 24 months
  The time interval from response to progression or death
Progression-free survival (PFS) | Until the end of the study or death, which may be up to 24 months
  The time interval from enrollment to progression or death
Overall survival (OS) | Until the end of the study or death, which may be up to 24 months
  The time interval from enrollment to death
Time to progression (TTP) | Until the end of the study or death, which may be up to 24 months
  the time interval from enrollment date to disease recurrence or progression except death
presence of genetic variation | at the time of enrollment
  homologous recombination deficiency [HRD] related genetic variation such as BRCA mutation
Number of of adverse events | Up to 24 months from the start of the intervention
  The investigator should review the measurement, examination, and assessment results of vital signs, physical examination, laboratory tests, ECG, etc. performed for the safety assessment, and assess and record the clinical significance of abnormal results. Any clinically significant abnormal findings (medical condition or abnormal values) should be collected as AEs.

CONTACTS AND LOCATIONS:
Overall Officials: Hee Seung Kim, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Suh DH, Chang SJ, Song T, Lee S, Kang WD, Lee SJ, Roh JW, Joo WD, Yoon JH, Jeong DH, Kim HS, Lee SJ, Ji YI, Kim HJ, Lee JW, Kim JW, Bae DS. Practice guidelines for management of ovarian cancer in Korea: a Korean Society of Gynecologic Oncology Consensus Statement. J Gynecol Oncol. 2018 Jul;29(4):e56. doi: 10.3802/jgo.2018.29.e56. Epub 2018 Mar 10. PMID 29770626
- [Background] Stover EH, Konstantinopoulos PA, Matulonis UA, Swisher EM. Biomarkers of Response and Resistance to DNA Repair Targeted Therapies. Clin Cancer Res. 2016 Dec 1;22(23):5651-5660. doi: 10.1158/1078-0432.CCR-16-0247. Epub 2016 Sep 27. PMID 27678458
- [Background] Gadducci A, Guarneri V, Peccatori FA, Ronzino G, Scandurra G, Zamagni C, Zola P, Salutari V. Current strategies for the targeted treatment of high-grade serous epithelial ovarian cancer and relevance of BRCA mutational status. J Ovarian Res. 2019 Jan 28;12(1):9. doi: 10.1186/s13048-019-0484-6. PMID 30691488
- [Background] Scambia G, Ferrandina G. A turning point in the fight against ovarian cancer? Lancet Oncol. 2018 Feb;19(2):154-156. doi: 10.1016/S1470-2045(18)30005-6. Epub 2018 Jan 18. No abstract available. PMID 29361471
- [Background] Obeidat B, Latimer J, Crawford R. Can optimal primary cytoreduction be predicted in advanced stage epithelial ovarian cancer? Role of preoperative serum CA-125 level. Gynecol Obstet Invest. 2004;57(3):153-6. doi: 10.1159/000076236. Epub 2004 Jan 15. PMID 14726621
- [Background] Smith J, Tho LM, Xu N, Gillespie DA. The ATM-Chk2 and ATR-Chk1 pathways in DNA damage signaling and cancer. Adv Cancer Res. 2010;108:73-112. doi: 10.1016/B978-0-12-380888-2.00003-0. PMID 21034966
- [Background] Jung KW, Won YJ, Kong HJ, Lee ES. Cancer Statistics in Korea: Incidence, Mortality, Survival, and Prevalence in 2016. Cancer Res Treat. 2019 Apr;51(2):417-430. doi: 10.4143/crt.2019.138. Epub 2019 Mar 18. PMID 30913865
- [Background] McGuire WP, Hoskins WJ, Brady MF, Kucera PR, Partridge EE, Look KY, Clarke-Pearson DL, Davidson M. Cyclophosphamide and cisplatin compared with paclitaxel and cisplatin in patients with stage III and stage IV ovarian cancer. N Engl J Med. 1996 Jan 4;334(1):1-6. doi: 10.1056/NEJM199601043340101. PMID 7494563
- [Derived] Park SJ, Chang SJ, Suh DH, Kong TW, Song H, Kim TH, Kim JW, Kim HS, Lee SJ. A phase IA dose-escalation study of PHI-101, a new checkpoint kinase 2 inhibitor, for platinum-resistant recurrent ovarian cancer. BMC Cancer. 2022 Jan 3;22(1):28. doi: 10.1186/s12885-021-09138-z. PMID 34980026